CLINICAL TRIAL: NCT07390214
Title: REFOCUS-AF - "RepEat Ablation With AFFERA vs. COntact Force-Guided RF Catheters for Optimal OUtcomes in Symptomatic AF".
Acronym: REFOCUS-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study Protocol Version 1.3
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation - Symptomatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CF-guided RFC: Re-PVI and substrate modification of low voltage areas (Experimental): Patient get intervention via Contact force guided radiofrequency ablation
  Interventions: Procedure: CF-guided RFC: Re-PVI and substrate modification of low voltage areas
- Dual Energy ablation with RF/PFA: Re-PVI and substrate modification of low voltage ath (Experimental): Patient will get Intervenstion via Large footprint PFA/RFC catheter (Sphere 9)
  Interventions: Procedure: Dual Energy ablation with RF/PFA: Re-PVI and substrate modification of low voltage areas

INTERVENTIONS:
Procedure: Dual Energy ablation with RF/PFA: Re-PVI and substrate modification of low voltage areas — Re-PVI
  Arms: Dual Energy ablation with RF/PFA: Re-PVI and substrate modification of low voltage ath
Procedure: CF-guided RFC: Re-PVI and substrate modification of low voltage areas — Re-PVI
  Arms: CF-guided RFC: Re-PVI and substrate modification of low voltage areas

SUMMARY:
This is a prospective, randomized (1:1), pilot study enrolling 200 patients with symptomatic atrial fibrillation or atrial tachycardia (AF/AT) recurrence requiring repeat ablation following a single prior PVI procedure for AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic non-valvular AF or AT recurrences despite of one previous PVI (+/- cavotricuspid isthmus ablation) catheter ablation for AF.

Age 18-85 years Willing and able to comply with the study protocol Willing and able to operate a device for rhythm monitoring

Exclusion Criteria:

* Patients with contraindications to catheter ablation or inability to provide informed consent Patients who underwent PVI + (ablation of additional RA/LA substrates/areas) Patients who did not undergo PVI before Patients who underwent more than one prior PVI/Re-PVI Patients with left atrial size > 55mm Patients with longstanding persistent AF > 12 months duration Prior surgical AF ablation Contraindications for repeat ablation Prior implantable loop recorder History of mitral valve surgery Severe mitral valve regurgitation Inability to be treated with oral anticoagulation Presence of intracardiac thrombi Chronic obstructive pulmonary disease or Asthma treated with long acting bronchodilatators Obstructive sleep apnea syndrome requiring CPAP mask ventilation Pregnancy Participation in other clinical studies Unwilling to follow the study protocol and to attend follow-up visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | Within the study duration of 1 Year
  Complete re-pulmonary vein isolation (re-PVI), Bidirectional conduction block across linear lesions, Complete substrate elimination (defined as: voltage abatement and/or loss of capture).

CONTACTS AND LOCATIONS:
Overall Officials: Julian Chun, Professor, Principal Investigator — MVZ CCB Germany
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, 60431, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided